CLINICAL TRIAL: NCT06337812
Title: Fiber Supplementation to Increase Short Chain Fatty Acid Production in Patients With Type II Diabetes and Heart Failure With Preserved Ejection Fraction - the FERMENT HFpEF Trial
Brief Title: Fiber Supplementation in Heart Failure With Preserved Ejection Fraction (HFpEF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Scott L. Hummel, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00240473
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Type2diabetes; Heart Failure With Preserved Ejection Fraction
Keywords: Fiber Supplementation; Potato Starch; Gut microbiome; Resistant starch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Potato starch supplement (Experimental): Participants will take the supplement for approximately 4 weeks.
  Interventions: Dietary Supplement: Potato Starch

INTERVENTIONS:
Dietary Supplement: Potato Starch — Participants will consume 10 grams (1/2 a packet) of Bob's Red Mill Potato Starch twice a day for the first 7 days and then increase to 20 grams (full packet) of potato starch for approximately 3 weeks. Potato starch can be mixed into cold food or beverage for consumption.
  In addition, participants will have evaluations and provide blood and stool samples during the study.

SUMMARY:
The study team is studying how increasing dietary fiber, specifically through adding potato starch to participant's diet, may impact the species of bacteria in participant's gut microbiome. The study team also wants to understand if adding potato starch to participant's diet helps these bacteria make more short chain fatty acids, a byproduct the team thinks may benefit participant's health.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed clinical diagnosis of stable HFpEF on maximally tolerated Heart Failure (HF) medical regimen (without changes in dosage in the prior month)
* Left ventricular ejection fraction of >50% documented in the prior 12 months
* A confirmed clinical diagnosis of Type II diabetes (T2DM) with glycated hemoglobin <10% without changes in medical regimen in the past month.

Exclusion Criteria:

* Current usage of pre- or probiotic usage
* Antibiotic usage in the past 6 months
* Current participation in another interventional clinical trial
* History of potato allergy or potato starch allergy, inflammatory bowel syndrome, inflammatory bowel disease, bowel resection, Roux-en-Y gastric bypass surgery, celiac disease, Crohn's disease, or colorectal cancer
* Hypoglycemic episode with blood glucose 70 milligrams per deciliter (mg/dL) within the last month
* Stage IV-V chronic kidney disease
* Pregnancy (self-reported)
* Comorbidity limiting survival to < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Short Chain Fatty Acid (SCFA) butyrate levels - stool | Baseline, approximately 4 weeks
  Stool will be analyzed.
Changes in Short Chain Fatty Acid (SCFA) butyrate levels - plasma | Baseline, approximately 4 weeks
  Plasma samples will be analyzed.
Changes in propionate levels - stool | Baseline, approximately 4 weeks
  Stool will be analyzed.
Changes in propionate levels- plasma | Baseline, approximately 4 weeks
  Plasma samples will be analyzed.
Changes in acetate levels- stool | Baseline, approximately 4 weeks
  Stool will be analyzed.
Changes in acetate levels- plasma | Baseline, approximately 4 weeks
  Plasma samples will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hummel, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No